CLINICAL TRIAL: NCT04335175
Title: Sensory Symptoms in Tourette Syndrome and Obsessive-Compulsive Disorder
Acronym: SenST-Plus
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Isaacs, Assistant Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: 200502
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Tourette Syndrome; Obsessive-Compulsive Disorder; Sensory Disorders
Keywords: sensory dysregulation; sensory gating dysfunction; tic; obsessive compulsive; sensory symptom
MeSH Terms: conditions — Tourette Syndrome; Obsessive-Compulsive Disorder; Sensation Disorders; Tics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tourette Syndrome: Individuals previously diagnosed with Tourette syndrome (TS). Participants must be 18 years of age or older.
  Interventions: Other: None - observational study
- Obsessive Compulsive Disorder: Individuals previously diagnosed with obsessive compulsive disorder (OCD). Participants must be 18 years of age or older.
  Interventions: Other: None - observational study
- Healthy Controls: Individuals with no past or current neurologic or psychiatric illness. Participants must be 18 years of age or older.
  Interventions: Other: None - observational study

INTERVENTIONS:
Other: None - observational study — None - observational study

SUMMARY:
This study seeks to address two key questions related to sensory dysregulation in Tourette syndrome (TS) and obsessive compulsive disorder (OCD): 1) Is sensory dysregulation in OCD clinically distinct from that in TS? 2) To what extent does sensory dysregulation affect QOL in each of these disorders? Patients with TS, patients with OCD, and healthy controls will complete an online battery of validated questionnaires assessing sensory dysregulation, psychiatric symptoms, and quality of life.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a neurodevelopmental disorder affecting 1% of school-aged children, with one-third of patients suffering persistent tics into adulthood. Obsessive-compulsive disorder (OCD) is a common comorbidity with TS. Individuals with either TS or OCD frequently exhibit sensory dysregulation, manifesting as heightened awareness of internal and external stimuli. For patients with OCD, sensory dysregulation has been linked to obsessive-compulsive symptoms and is an important consideration in treatment strategies. Sensory dysregulation remains largely unexplored in TS, but preliminary data suggests it is dissociable from tics, linked with obsessive-compulsive symptoms, and associated with poorer quality of life (QOL). This study seeks to address two key questions related to sensory dysregulation in TS and OCD: 1) Is sensory dysregulation in OCD clinically distinct from that in TS? 2) To what extent does sensory dysregulation affect QOL in each of these disorders? To do so, we will recruit patients with TS, patients with OCD, and healthy controls to complete an online battery of validated questionnaires assessing sensory dysregulation, psychiatric symptoms, and QOL. Addressing these knowledge gaps will enhance our understanding of bothersome sensory symptoms in TS and OCD, shed light on clinical overlap and/or distinctions between these commonly co-occurring psychiatric diagnoses, and clarify QOL impact and the potential need for more direct targeting of these symptoms.

ELIGIBILITY:
Inclusion criteria for the patient groups:

* age 18 years or older
* previous diagnosis of Tourette syndrome and/or obsessive compulsive disorder

Exclusion criteria for the patient groups:

- none

Inclusion criteria for healthy controls includes:

- 18 years of age or older

Exclusion criteria for the patient groups:

- history of any neurologic or psychiatric diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years of age or older with Tourette syndrome and/or obsessive compulsive disorder.
  Individuals 18 years of age or older with no neurologic or psychiatric diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Sensory Gating Inventory | Day 1
  36-item, validated self-report questionnaire assessing sensory gating symptoms, with score range 0-216. Higher scores indicate greater sensory gating impairment.

SECONDARY OUTCOMES:
Dimensional Obsessive Compulsive Scale | Day 1
  20-item, validated self-report questionnaire assessing obsessive compulsive symptoms, with score range 0-80. Higher scores indicate more severe obsessive compulsive symptoms.
Adult Attention Deficit Hyperactivity Disorder Self-Report Screening Scale | Day 1
  6-item, validated self-report questionnaire assessing inattention and hyperactivity symptoms, with raw score range from 0-24. Higher scores indicate greater ADHD symptoms.
Generalized Anxiety Disorder-7 Scale | Day 1
  7-item, validated self-report questionnaire assessing anxiety symptoms, with score range from 0-21. Higher scores indicate more severe anxiety.
Patient Health Questionnaire-9 Scale | Day 1
  9-item, validated self-report questionnaire assessing depression symptoms, with score range from 0-27. Higher scores indicate more severe depression.
Premonitory Urge to Tic Scale (for Tourette syndrome patients only) | Day 1
  10-item, validated self-report questionnaire assessing premonitory urge symptoms, with score range from 9-36. Higher scores indicate more severe premonitory urge prior to tics.
Adult Tic Questionnaire (for Tourette syndrome patients only) | Day 1
  27-item, validated self-report questionnaire assessing frequency and severity of tics, with score range from 54-216. Higher scores indicate greater tic burden.
WHO Quality of Life - BREF | Day 1
  26-item, validated self-report questionnaire assessing 4 domains of health: physical, psychological, social, and environmental.
  54-216. Higher scores indicate greater tic burden. Scores range from 0-100 within each domain. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: David Isaacs, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified participant data collected, study protocol, statistical analysis plan, and informed consent documents will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to david.a.isaacs@vumc.org. To gain access, data requestors will need to sign a data access agreement.